CLINICAL TRIAL: NCT06717776
Title: Effects of Compensation-Based Problem-Solving Therapy on Occupational Performance, Self Efficacy, Participation and Quality of Life After Stroke: A Randomized Controlled Trial
Brief Title: Effects of Compensation-Based Problem Solving Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Kaya Ozturk, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HÜ-OT-LKO-01
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: stroke; compensation; self-efficacy; problem solving; participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two groups with an intervention group and a control group
Who Masked: Outcomes Assessor
Masking Description: The therapist who conducted the assessment tests was unaware of the participants' group assignments (interventon or control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (intervention group) (Active Comparator): The intervention group received both compensation-bocused problem-solving therapy and standard rehabilitation services.
  Standard Rehabilitation:The program allows individuals to utilize the physiotherapy and occupational therapy units on a weekly basis, with access available on weekdays.
  Compensation Based Problem Solving Therapy (CFPS) is an approach based on the occupational adaptation model. It entails the implementation of compensatory strategies with the objective of enhancing the performance of both extremities in activities of daily living.
  Interventions: Behavioral: Compensation Based Problem Solving Therapy; Behavioral: standard rehabilitation
- Plasebo (control group) (Active Comparator): The control group received standard rehabilitation services.
  Standard Rehabilitation:The program allows individuals to utilize the physiotherapy and occupational therapy units on a weekly basis, with access available on weekdays.
  Interventions: Behavioral: standard rehabilitation

INTERVENTIONS:
Behavioral: Compensation Based Problem Solving Therapy — Compensation-Based Problem Solving Therapy (CB-PST) is a therapeutic approach based on the occupational adaptation model. It entails the implementation of compensatory strategies with the objective of enhancing the performance of both extremities in daily life activities. The therapy encompasses the implementation of problem-solving training.
  The occupational problem is defined.
  The development of compensation-focused strategies is based on the "personal factors" and "occupational environment" identified as relevant to the problematic occupation, as determined according to the principles of the occupational adaptation model.
  Once a compensatory strategy has been selected, the next step is to apply it and evaluate its efficacy, with the expectation that an "adaptive response" will be observed, and that the resulting adaptation will be reflected in improved occupational performance, as guided by the occupational adaptation model.
  Arms: Aspirin (intervention group)
Behavioral: standard rehabilitation — The standard rehabilitation program is provided to all individuals in the inpatient service on an equal basis. The program allows individuals to utilize the physiotherapy and occupational therapy units on a weekly basis, with access available on weekdays. These units are staffed by physiotherapists and occupational therapists. All individuals included in the study received the same service from the same therapists at the same times in a homogeneous manner. All individuals received physiotherapy, electrotherapy, and hydrotherapy as part of this service. In the physiotherapy unit, the first intervention was 25 minutes of electrotherapy for the upper extremity. This was followed by 40 minutes of physiotherapy exercises, conducted with the assistance of a physiotherapist. The final component of the physiotherapy unit programme was 15 minutes of hydrotherapy. In the occupational therapy unit, a standard 40-minute occupa

SUMMARY:
The aim of the study was to develop a Compensation-Based Problem-Solving Therapy and to examine its effects on occupational performance, participation, self-efficacy, and quality of life in individuals with stroke.

DETAILED DESCRIPTION:
The study was designed as a randomized controlled trial. A simple randomization method was employed to randomly assign individuals to two groups (intervention and control groups). A simple randomization method was employed, whereby the intervention and control group papers were selected from a closed envelope. Following the initial evaluation of each participant, one of the papers bearing the designation "intervention" or "control" was selected at random. This decision determined whether the individual would be included in the intervention or control group. The study was conducted in the occupational therapy department of the physical therapy and rehabilitation clinic of Etlik City Hospital. The study was approved by the Ethics Committee of Etlik City Hospital on May 17, 2023, and was assigned the code AEŞH-EK1-2023-176. Following approval from the ethics committee, the Compensation-Based Problem Solving Training (CBPST) was developed. The training program was developed in accordance with the tenets of the Occupational Adaptation Model. All subsequent steps were conducted in accordance with the aforementioned model. The adaptive response, as outlined in the model, encompasses the occupational adaptation that is anticipated to occur at the conclusion of the training program. The therapy was then trialled with a pilot group of five individuals, with the aim of refining the content. Subsequently, the final iteration of the training program was established. All individuals included in the study signed a consent form indicating their willingness to participate. This was completed at the outset of the study. All individuals were provided with a standard rehabilitation program comprising five days a week (40 minutes) of routine therapy. In addition to this, the intervention group received CBPST in the form of five days a week (20 minutes) sessions. The evaluations completed at the beginning of the training were repeated one month later.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ischemic stroke due to middle cerebral artery lesion 18-64 years of age Stroke time between 3-12 months Scoring 24 and above on the Standardized Mini Mental Test Scoring 16 and below on the NIH Stroke Scale Receiving service in the inpatient service at Etlik City Hospital

Exclusion Criteria:

* Having any psychiatric or neurological disease that may affect the study Individuals whose affected hand is not their dominant hand Individuals who tend to neglect their affected hand

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | 1 month
  The Canadian Occupational Performance Measure (COPM) is a measurement tool that is specific to the individual and is used to evaluate the performance and satisfaction of individuals in their activities of daily living. The COPM employs a person-centered approach, encompasses a comprehensive scope, and assesses performance and satisfaction. The tool includes the following components: problem definition, prioritization, scoring, goal setting, and re-evaluation. The COPM comprises three domains of occupational performance: self-care, work and productive activities, and leisure time activities. The individual's desired occupations within these areas are identified and assigned a score between 1 and 10. Subsequently, the five most significant occupations are identified from the aforementioned list and performance and satisfaction scores are assigned a value between 1 and 10. The total performance and total satisfaction levels of these occupations are then recorded. Additionally, the total

SECONDARY OUTCOMES:
The Stroke Specific Quality of Life Scale (SSQLS) | 1 month
  The Stroke Specific Quality of Life Scale (SSQLS) is a measurement tool developed for the purpose of evaluating the quality of life of individuals who have experienced a stroke. This scale is employed to ascertain the impact of stroke on the physical, emotional, and social well-being of the individual, thereby informing the formulation of treatment and intervention plans that align with these effects. The scale has the advantages of being a stroke-specific tool, comprehensive, and sensitive to the patient. The scale comprises 12 domains and 49 items. The aforementioned areas encompass the following domains: energy, family roles, movement, emotions, personal care, social roles, communication, vision, thinking, upper extremity functions, pain, work and productivity. The item numbers in these areas vary. However, each area is scored using a Likert-type scale, with scores ranging from 1 (indicating a high level of dissatisfaction) to 5 (indicating a high level of satisfaction). Subsequent
Daily Living Self Efficacy Scale | 1 month
  It is a tool used to evaluate one's own efficacy in everyday activities. This scale assesses an individual's capacity to fulfill specific roles and responsibilities, providing an insight into their intrinsic capability. The concept of self-efficacy is comprised of two sub-categories: social and everyday. The psychosocial sub-category encompasses eight items, while the activies of daily living sub-category encompasses four items, for a total of 12 items. A rating system is in use, with a scale of 0 to 100. A higher score is indicative of a higher level of self-efficacy.
Participation Scale | 1 month
  It is a measurement tool utilized to assess the extent of individual participation in social activities and the constraints they encounter in this participation. The scale was developed with the specific purpose of measuring social isolation and understanding the capacity of individuals to fulfill their roles in society. The P-Scale is typically employed to assess the level of participation of individuals coping with chronic illnesses, physical disabilities, mental health concerns, or social disadvantages within society. The scale comprises 18 items, with responses scored on a Likert scale from 1 (no problems) to 5 (severe participation restrictions). A high score indicates a significant limitation in the individual's capacity to engage in social activities. The scale offers several advantages, including cultural flexibility, straightforward administration, individualized assessment, and sensitivity to the specific circumstances of the individual being evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effectiveness of problem solving therapy for stroke patients: study protocol for a pragmatic randomized controlled trial — https://link.springer.com/article/10.1186/1471-2377-13-67